CLINICAL TRIAL: NCT07119515
Title: A Randomized Controlled Trial Comparing Teletherapy and In-Person Third-Wave CBT for Generalized Anxiety Disorders
Brief Title: Teletherapy vs. In-Person Cognitive Behavioral Therapy for Generalized Anxiety Disorder
Acronym: TIPCBT-GAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Collaborators: Allied Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Imaan Sabeeh, MS Scholar , Department of Applied Psychology, GCUF, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCUF-IRB-585-2025
Record Dates: First submitted 2025-04-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Generalized Anxiety Disorder
Keywords: Teletherapy; In-person therapy; Cognitive behavioral therapy (CBT); Generalized anxiety disorder (GAD); Randomized controlled trial (RCT); Mental health accessibility; Anxiety disorders; Pakistan; Therapeutic alliance; Third-wave CBT; Remote mental health services
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teletherapy (Experimental)
  Interventions: Behavioral: Third-Wave CBT via Teletherapy
- In-Person therapy (Active Comparator)
  Interventions: Behavioral: Third-Wave CBT In-Person

INTERVENTIONS:
Behavioral: Third-Wave CBT via Teletherapy — Twelve weekly 40-minute remote sessions via video conferencing, including mindfulness, behavioral activation, and exposure therapy.
  Arms: Teletherapy
Behavioral: Third-Wave CBT In-Person — Twelve weekly 40-minute face-to-face sessions with identical third-wave CBT content.
  Arms: In-Person therapy

SUMMARY:
The goal of this randomized controlled trial is to compare the clinical efficacy of teletherapy versus in-person third-wave cognitive behavioral therapy (CBT) in treating generalized anxiety disorder (GAD) among young individuals aged 18-45 years in Pakistan. The main questions it aims to answer are:

* Is teletherapy as effective as in-person therapy in reducing anxiety symptoms and stress?
* Do therapeutic alliance, treatment adherence, and social support influence treatment outcomes differently across delivery methods? Researchers will compare the teletherapy group (remote sessions via digital platforms) and the in-person therapy group (face-to-face sessions) to evaluate differences in symptom reduction, general health improvement, and moderating factors like therapeutic alliance.

Participants will:

* Undergo a 8-week intervention with weekly structured third-wave CBT sessions.
* Complete assessments at baseline, post-intervention, and follow-up using validated scales (e.g., Generalized Anxiety Disorder-7 [GAD-7], Hamilton Anxiety Rating Scale [HAM-A]).
* Engage in modules including mindfulness, behavioral activation, and exposure therapy, adapted for their assigned delivery method.

This study aims to address gaps in mental health accessibility in Pakistan by evaluating whether teletherapy can serve as a viable alternative to traditional in-person care.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) compares the efficacy of teletherapy versus traditional in-person delivery of third-wave cognitive behavioral therapy (CBT) for treating generalized anxiety disorder (GAD) among adults (aged 18-45 years) in Pakistan. Conducted at Allied Hospital II, Faisalabad, the study will randomize eligible participants(diagnosed via Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision [DSM-5-TR] criteria) into two parallel arms: (1) a teletherapy group receiving 12 weekly sessions via secure video conferencing, and (2) an in-person group attending face-to-face sessions with identical content. Both interventions will follow a standardized third-wave CBT protocol integrating mindfulness, acceptance, and behavioral strategies. Primary outcomes include changes in anxiety severity (measured by Hamilton Anxiety Rating Scale [HAM-A] and Generalized Anxiety Disorder-7 [GAD-7]) and depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]). Secondary outcomes assess perceived stress (Perceived Stress Scale [PSS]), work and social adjustment (Work and Social Adjustment Scale [WSAS]) and therapeutic alliance (Working Alliance Inventory [WAI]). Assessments will occur at baseline, post-intervention, and follow-up. The study aims to address critical gaps in mental healthcare accessibility in resource-limited settings by evaluating whether teletherapy can achieve comparable outcomes to in-person therapy. Ethical approval will be obtained from GCUF's Institutional Review Board (IRB), and the trial adheres to Consolidated Standards of Reporting Trials (CONSORT) guidelines. Results may inform policy decisions to expand remote mental health services in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18-≤45 years -meeting the diagnostic criteria according to DSM-5 TR -ability to understand and read English -ability to use digital technology and having access to the Internet -signed an informed consent form

Exclusion Criteria:

* the presence of risk of suicide and self-destructive behaviors -presence of another severe mental disorder (i.e., substance abuse, psychotic disorder, or bipolar disorder) -presence of severe personality disorder -presence of a medical condition whose severity or characteristics prevent participation in treatment -receiving another psychological treatment during the study
* an increase or change in medication during the study period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | 3 Months
  A clinician-rated scale assessing anxiety severity. Range: 0-56 (higher scores indicate worse outcomes).
Generalized Anxiety Disorder-7 (GAD-7) | 3 Months
  A 7-item self-report questionnaire measuring anxiety severity. Range: 0-21 (higher scores indicate worse outcomes).
Patient Health Questionnaire-9 (PHQ-9) | 3 Months
  A 9-item self-report tool for assessing depressive symptoms. Range: 0-27 (higher scores indicate worse outcomes).

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 3 Months
  A 10-item self-report measure evaluating perceived stress. Range: 0-40 (higher scores indicate worse outcomes).
Work and Social Adjustment Scale (WSAS) | 3 Months
  A 5-item self-report measure assessing functional impairment in work and social domains. Range: 0-40 (higher scores indicate worse outcomes).
Working Alliance Inventory (WAI) | 3 Months
  A 12-item scale measuring therapeutic alliance between client and therapist. Range: 12-84 (higher scores indicate better outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Imaan Sabeeh, MS Scholar, Principal Investigator — Government College University Faisalabad
Locations (1):
- Allied Hospital II, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request to qualified researchers. Data will include baseline characteristics, outcome measures, treatment adherence metrics, and supporting documents such as the study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available six months post-publication
Access Criteria: Access will be granted to researchers affiliated with academic institutions, non-profit organizations, or governmental agencies for non-commercial research purposes. De-identified IPD (demographics, clinical outcomes, treatment data) and supporting documents (protocol, statistical analysis plan, informed consent template) can be assessed. Data will be accessible after publication of the primary study results.
URL: https://osf.io/wscnb/